CLINICAL TRIAL: NCT03877133
Title: Association of Intraoperative Renal Regional Oxygen Saturation and Acute Kidney Injury After Living Donor Liver Transplantation
Brief Title: Association of Intraoperative Renal Regional Oxygen Saturation and Acute Kidney Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Associate Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1901-087-100
Record Dates: First submitted 2019-03-08; First posted 2019-03-15 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Liver Transplant; Complications; Renal Injury
Keywords: Near-infrared spectroscopy; Renal regional oxygen saturation; Living donor liver transplantation; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: A prospective, single group, observational study
Masking Description: Does not need masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regional oxygen saturation group (Other): Near-infrared spectroscopy application to the skin near the kidney
  Interventions: Device: Near-infrared spectroscopy

INTERVENTIONS:
Device: Near-infrared spectroscopy — Regional oxygen saturation probe is applied to the skin near the kidney bilaterally and is connected to the regional oxygen saturation monitor.

SUMMARY:
This study is a prospective observational study of a single cohort of the patients who will undergo a scheduled living donor liver transplantation.

The investigators attempt to evaluate the association of intraoperative renal regional oxygen saturation and acute kidney injury in patients undergoing living donor liver transplantation. Near-infrared spectroscopy sensor will be attached to the skin near bilateral kidney areas in all patients and renal regional oxygen saturation will be monitored during the operation. Renal regional oxygen saturation (rSO2) of the patients who developed acute kidney injury postoperatively will be compared with rSO2 of the patients who did not.

DETAILED DESCRIPTION:
Acute kidney injury is a frequent complication after liver transplantation, which is related to poor prognosis and longer hospital stay. There is no sensitive or specific marker for predicting postoperative acute kidney injury, although studies of the biomarkers have shown promising results.

Near-infrared spectroscopy is a non-invasive and real-time monitoring device for regional oxygen saturation measurement. Previous studies revealed that it could be applied to the skin near the kidney and be used to monitor renal regional oxygen saturation.

Therefore, in this study, the investigators will apply near-infrared spectroscopy around kidney area to measure real-time renal regional oxygen saturation during liver transplantation surgery and investigate the association between the intraoperative renal regional oxygen saturation and the development of post-transplant acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled to undergo elective living donor liver transplantation
* Patients who provided written informed consent

Exclusion Criteria:

* Missing preoperative serum creatinine value
* Underlying kidney disease, such as hepatorenal syndrome, chronic kidney disease
* History of unilateral or bilateral nephrectomy
* Patients who died within 48 hours immediately after surgery
* Any skin problem at the attachment site of regional oxygen saturation probe

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury | Within 7 days after surgery
  Acute kidney injury defined by the Kidney Disease Improving Global Outcomes (KDIGO) criteria using postoperative serum creatinine

SECONDARY OUTCOMES:
Length of hospital stay | Within 30 days after surgery
  Length of hospital stay
Nadir oxygen delivery during the surgery | Within average 8 hours after anesthesia induction during the transplantation surgery
  Nadir oxygen delivery calculated by the cardiac output and arterial oxygen content
Area under the curve of oxygen delivery during the surgery | Within average 8 hours after anesthesia induction during the transplantation surgery
  Area under the curve of oxygen delivery calculated by the cardiac output and arterial oxygen content
Early allograft dysfunction | on the postoperative 7th day after liver transplantation
  Early allograft dysfunction diagnosed by one or more of the following variables: (1) bilirubin > 10 mg/dL on postoperative day 7; (2) prothrombin time: international normalized ratio > 1.6 on postoperative day 7; (3) aminotransferase level (alanine aminotransferase or aspartate aminotransferase > 2000 IU/ml within the first 7 postoperative days.
In-hospital mortality | Within 30 days after surgery
  In-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No